CLINICAL TRIAL: NCT01802983
Title: Key Technology Research of the Comprehensive Treatment of Multiple Organ Dysfunction Syndrome
Brief Title: The Prognostic Assessment of Extubation in Aged Patients With Multiple Organ Dysfunction Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Kun Xiao, Key Technology Research of the comprehensive treatment of Multiple organ dysfunction syndrome, Chinese PLA General Hospital
Other Study IDs: 2013670808
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Organ Dysfunction Syndrome
Keywords: Aged; Multiple organ failure; Extubation; Prognosis; MODS; invasive mechanical ventilation
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The multiple organ dysfunction syndrome (MODS) has remained the major factor contributing to prolongation of intensive and mortality. It is reported that the mortality rates have varied between 20% and 100%, depending on number, severity, duration, type and combination, and definition of dysfunction. In our study, the investigators explore some comprehensive treatment technology to improved outcomes of MODS patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 60 years old;
* presence of altered organ function in an acutely ill patient such that homeostasis cannot be maintained without intervention;
* have trachea intubation after admitting to intensive care unit within 24 hours.

Exclusion Criteria:

* end stage multiple organ failure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between Jan 2009 and May 2013 in the Respiratory Intensive Care Unit(RICU),Surgical Intensive Care Unit(SICU) and Emergency Intensive Care Unit(EICU).
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
the prognostic assessment of aged patients with MODS | 28 days
  According to the outcomes of 28-day,all the enrolled patients were divided into survival group and death group, clinical datum of which were collected and analysed. And then these prognosis were evaluated with the current scoring systems [(Acute Physiology and Chronic Health EvaluationⅡ(APACHEⅡ, APACHE Ⅲ), Sample Acute Physiological score(SAPSⅡ), Multiple Organ Dysfunction score(MODS)], the predictive power of which were compared by receiver operating characteristic(ROC) curve. Finally, a binary logistic regression analysis was performed to evaluate the concerning prognostic factors of MODSE.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xiao K, Su L, Han B, Guo C, Feng L, Jiang Z, Wang H, Lin Y, Jia Y, She D, Xie L. Prognosis and weaning of elderly multiple organ dysfunction syndrome patients with invasive mechanical ventilation. Chin Med J (Engl). 2014;127(1):11-7. PMID 24384417